CLINICAL TRIAL: NCT07167589
Title: Capsule Bag Performance of a Novel Single-piece Acrylic IOL HOYA AF-1 NY-60
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Viros_HOYA
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2010-04

CONDITIONS: Cataract Surgery, Single-piece IOL, Microincisional IOL
MeSH Terms: interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HOYA acrylic single-piece IOL (HOYA AF-1 NY-60) (Other)
  Interventions: Procedure: Cataract surgery with implantation of a single-piece microincisional IOL

INTERVENTIONS:
Procedure: Cataract surgery with implantation of a single-piece microincisional IOL

SUMMARY:
During the past decades, cataract surgery underwent tremendous change and modernisation resulting in today's small incision, phacoemulsification surgery and a safe technique with a short rehabilitation time for the patient.

In this study the capsule performance and stability of a new one-piece microincisional hydrophobic acrylic IOL (HOYA AF-1 NY-60) should be assessed in subgroups of normal, short and long eyes. The IOL has a sharp optic edge design to inhibit PCO formation. Hypothesis: The novel haptic design is supposed to avoid tension folds in capsule bag, allow for a longer contact length of haptic with capsule equator, ensure rotational stability as well as good centration of the optic.

ELIGIBILITY:
Inclusion Criteria:

* Age-related cataract
* Age 21 and older
* Visual Acuity > 0.05
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant

Exclusion Criteria:

* Relevant other ophthalmic diseases especially those that may compromise capsule bag integrity or zonule stability (such as pseudoexfoliation syndrome, Marfan's syndrome, etc.)
* Preceding ocular surgery or trauma
* In case of pregnancy (pregnancy test will be taken preoperatively in women of reproductive age)

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-02-01 (Actual); Primary Completion 2013-05-01 (Actual); Study Completion 2013-12-01 (Actual)

PRIMARY OUTCOMES:
Anterior chamber depth | 4 times, each 5 minutes during procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Vienna Institute for Research in Ocular Surgery, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided